CLINICAL TRIAL: NCT02989857
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-controlled Study of AG-120 in Previously-treated Subjects With Nonresectable or Metastatic Cholangiocarcinoma With an IDH1 Mutation
Brief Title: Study of AG-120 in Previously Treated Advanced Cholangiocarcinoma With IDH1 Mutations (ClarIDHy)
Acronym: ClarIDHy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG120-C-005
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Advanced Cholangiocarcinoma; Metastatic Cholangiocarcinoma
Keywords: IDH1
MeSH Terms: conditions — Cholangiocarcinoma | interventions — ivosidenib

STUDY DESIGN:
Intervention Model Description: Patients randomized in a 2:1 allocation (AG-120 vs Placebo)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AG-120 (Active Comparator): Participants received AG-120 500 mg, tablet, orally, once a day (QD) in each 28-day treatment cycle, until occurrence of disease progression, unacceptable toxicity, confirmed pregnancy, death, subject withdrawal, lost to follow-up, or the sponsor ended the study for up to approximately 45 months.
  Interventions: Drug: AG-120
- Placebo (Placebo Comparator): Participants received AG-120 matched placebo, orally, QD in each 28-day treatment cycle, until occurrence of disease progression, unacceptable toxicity, confirmed pregnancy, death, subject withdrawal, lost to follow-up or the sponsor ended the study for up to approximately 7 months. Participants who experienced disease progression and received placebo were allowed to cross over and receive AG-120.
  Interventions: Drug: Placebo
- After Cross over to AG-120 (Experimental): Participants who experienced disease progression and received placebo were allowed to cross over to receive AG-120 500 mg, tablet, orally, QD in each 28-day treatment cycle for up to approximately 32 months.
  Interventions: Drug: AG-120

INTERVENTIONS:
Drug: AG-120 — Tablet administered orally
  Other Names: Ivosidenib
  Arms: AG-120; After Cross over to AG-120
Drug: Placebo — Tablet administered orally
  Arms: Placebo

SUMMARY:
Study AG120-C-005 is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study of orally administered AG-120. Participants, all personnel involved in the evaluation of participants' response to treatment (e.g., Investigators, study coordinators, study pharmacists), and designated Sponsor team members will be blinded to study treatment. Participants are required to have a histologically-confirmed diagnosis of isocitrate dehydrogenase-1 (IDH1) gene-mutated cholangiocarcinoma that is not eligible for curative resection, transplantation, or ablative therapies prior to enrollment. IDH1 mutation testing will be performed at participating investigative sites. Participants must have progression of disease and have received at least 1 but not more than 2 prior treatment regimens for advanced disease (nonresectable or metastatic). All participants must have received either a gemcitabine or a 5 fluorouracil (5-FU) based chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age.
2. Have a histopathological diagnosis (fresh or banked tumor biopsy sample, preferably collected within the last 3 years) of nonresectable or metastatic cholangiocarcinoma and are not eligible for curative resection, transplantation, or ablative therapies.
3. Have documented IDH1 gene-mutated disease (from a fresh tumor biopsy or the most recent banked tumor tissue available) based on central laboratory testing (R132C/L/G/H/S mutation variants tested).
4. Have an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1
5. Have an expected survival of ≥3 months.
6. Have at least one evaluable and measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Participants who have received prior local therapy (including but not limited to embolization, chemoembolization, radiofrequency ablation, or radiation therapy) are eligible provided measurable disease falls outside of the treatment field or within the field and has shown ≥20% growth in size since post-treatment assessment.
7. Have documented disease progression following at least 1 and no more than 2 prior systemic regimens for advanced disease (nonresectable or metastatic). Participants must have received at least 1 gemcitabine- or 5-FU-containing regimen for advanced cholangiocarcinoma. Participants who have received systemic adjuvant chemotherapy will be permitted provided there is documented disease progression during or within 6 months of completing the therapy.

Exclusion criteria:

1. Received a prior IDH inhibitor.
2. Received systemic anticancer therapy or an investigational agent <2 weeks prior to Day 1 (washout from prior immune based anticancer therapy is 4 weeks). In addition, the first dose of study treatment should not occur before a period ≥5 half-lives of the investigational agent has elapsed.
3. Received radiotherapy to metastatic sites of disease <2 weeks prior to Day 1.
4. Underwent hepatic radiation, chemoembolization, and radiofrequency ablation <4 weeks prior to Day 1.
5. Have known symptomatic brain metastases requiring steroids. Participants with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and have radiographically stable disease for at least 3 months prior to study entry. Note: up to 10 mg per day of prednisone equivalent will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs Servier Pharmaceuticals LLC, Study Chair — Servier Pharmaceuticals, LLC
Locations (49):
- United States (26):
  - Mayo Cancer Center, Scottsdale, Arizona
  - City of Hope Cancer Center, Duarte, California
  - University of California, Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Mayo Cancer Center, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Cancer Center, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, SouthWestern, Dallas, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Carbone Cancer Center, Madison, Wisconsin
- France (4):
  - Universite de Franche-Comte, Besançon
  - Centre de Lutte Contre le Cancer (CLCC) - Institut Bergonie, Bordeaux
  - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer, Rennes
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Fondazione del Piemonte per l'Oncologia - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS Candiolo), Candiolo
  - Istituto Scientifico Universitario San Raffaele, Milan
  - Istituto Clinico Humanitas, Rozzano
- South Korea (6):
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul, St. Mary's Hospital, Seoul
  - National Cancer Center, Seoul
- Spain (5):
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
- United Kingdom (5):
  - St. James University Hospital, Leeds
  - Liverpool Cancer Center, Liverpool
  - University College London Hospitals, London
  - The Royal Free Hospital, London
  - The Christie NHS Foundation Trust, the Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Abou-Alfa GK, Macarulla T, Javle MM, Kelley RK, Lubner SJ, Adeva J, Cleary JM, Catenacci DV, Borad MJ, Bridgewater J, Harris WP, Murphy AG, Oh DY, Whisenant J, Lowery MA, Goyal L, Shroff RT, El-Khoueiry AB, Fan B, Wu B, Chamberlain CX, Jiang L, Gliser C, Pandya SS, Valle JW, Zhu AX. Ivosidenib in IDH1-mutant, chemotherapy-refractory cholangiocarcinoma (ClarIDHy): a multicentre, randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Jun;21(6):796-807. doi: 10.1016/S1470-2045(20)30157-1. Epub 2020 May 13. PMID 32416072
- [Derived] Valle JW, Abou-Alfa GK, Kelley RK, Lowery MA, Shroff RT, Bian Y, Saint-Hilary G, Liu H, Teng Z, Hua Z, Gliser C, Vogel A, Javle MM. Quantitative benefit-risk assessment of data from the phase III ClarIDHy study of ivosidenib versus placebo in patients with mIDH1 cholangiocarcinoma. ESMO Gastrointest Oncol. 2025 Apr 3;8:100159. doi: 10.1016/j.esmogo.2025.100159. eCollection 2025 Jun. PMID 41646284
- [Derived] Fan B, Abou-Alfa GK, Zhu AX, Pandya SS, Jia H, Yin F, Gliser C, Hua Z, Hossain M, Yang H. Pharmacokinetics/pharmacodynamics of ivosidenib in advanced IDH1-mutant cholangiocarcinoma: findings from the phase III ClarIDHy study. Cancer Chemother Pharmacol. 2024 May;93(5):471-479. doi: 10.1007/s00280-023-04633-5. Epub 2024 Jan 27. PMID 38278871
- [Derived] Zhu AX, Macarulla T, Javle MM, Kelley RK, Lubner SJ, Adeva J, Cleary JM, Catenacci DVT, Borad MJ, Bridgewater JA, Harris WP, Murphy AG, Oh DY, Whisenant JR, Lowery MA, Goyal L, Shroff RT, El-Khoueiry AB, Chamberlain CX, Aguado-Fraile E, Choe S, Wu B, Liu H, Gliser C, Pandya SS, Valle JW, Abou-Alfa GK. Final Overall Survival Efficacy Results of Ivosidenib for Patients With Advanced Cholangiocarcinoma With IDH1 Mutation: The Phase 3 Randomized Clinical ClarIDHy Trial. JAMA Oncol. 2021 Nov 1;7(11):1669-1677. doi: 10.1001/jamaoncol.2021.3836. PMID 34554208
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 49 study sites in France, Italy, Spain, South Korea, the United States, and the United Kingdom from 20 February 2017 to 17 May 2021.
Pre-assignment Details: The final analysis of progression-free survival (PFS) occurred once 131 PFS events had been determined by Investigator assessment. Two participants were randomized in the study after the data cutoff date (31 January 2019) for the final analysis of PFS.
Groups:
- AG-120: Participants received AG-120 500 mg, tablet, orally, once daily (QD) in each 28-day treatment cycle, until occurrence of disease progression, unacceptable toxicity, confirmed pregnancy, death, subject withdrawal, lost to follow-up, or the sponsor ended the study for up to approximately 45 months.
- After Crossover to AG-120: Participants who experienced disease progression and received placebo were allowed to cross over to receive AG-120 500 mg, tablet, orally, QD in each 28-day treatment cycle for up to approximately 32 months.
Period: Randomization Phase
Arm/Group | AG-120 | Placebo | After Crossover to AG-120
Started | 126 | 61 | 0
Completed | 123 (Completed = Participants who completed the protocol defined treatment.) | 59 (Completed = Participants who completed the protocol defined treatment.) | 0
Not Completed | 3 | 2 | 0
Not completed — Not Treated | 3 | 2 | 0
Period: Cross Over Phase
Arm/Group | AG-120 | Placebo | After Crossover to AG-120
Started | 0 | 0 | 43 (Participants who had experienced disease progression and received placebo were allowed to cross over to receive AG-120.)
Completed | 0 | 0 | 43 (Completed = Participants who completed the protocol defined treatment.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Set included all participants who were randomized, with the treatment group designated according to the randomization.
Groups:
- AG-120: Participants received AG-120 500 mg, tablet, orally, QD in each 28-day treatment cycle, until occurrence of disease progression, unacceptable toxicity, confirmed pregnancy, death, subject withdrawal, lost to follow-up, or the sponsor ended the study for up to approximately 45 months.
- Total: Total of all reporting groups
Arm/Group | AG-120 | Placebo | Total
Number analyzed (Participants) | 126 | 61 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.97) | 62.9 (10.38) | 61.1 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 37 | 119
  Male | 44 | 24 | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 7 | 2 | 9
  Ethnicity: Not Hispanic or Latino | 84 | 40 | 124
  Ethnicity: Not Reported | 0 | 2 | 2
  Ethnicity: Missing | 35 | 17 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 15 | 8 | 23
  Race: Black or African American | 1 | 1 | 2
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: White | 71 | 35 | 106
  Race: Other | 1 | 0 | 1
  Race: Not Reported | 1 | 0 | 1
  Race: Missing | 35 | 17 | 52

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Determined by the Independent Radiology Committee (IRC)
Description: PFS is defined as the time from date of randomization to the date of first documented disease progression as assessed by the IRC using Response Evaluation Criteria in Solid Tumors [RECIST] v1.1, or date of death due to any cause, whichever occurred first. Disease progression was defined as greater than or equal to (≥)20 percent (%) increase in sum of the diameter of target lesions, taking as reference the smallest sum diameter recorded since the treatment started. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm) or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization to the date of first documentation of disease progression or death due to any cause (Up to approximately 2 years)
Population: ITT set included all participants who were randomized, with the treatment group designated according to the randomization. Number analyzed is the number of participants with data available for analyses at the specified time point. Two participants were excluded from the analysis as they were randomized in the study after the data cutoff date (31 January 2019) for the analysis of PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 124 | 61
months | 2.7 [1.6 to 4.2] | 1.4 [1.4 to 1.6]
Statistical Analysis 1: Comparison: AG-120 vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — P-value was calculated from the one-sided stratified log-rank test; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.25 to 0.54] — Hazard ratio was calculated from stratified Cox regression model with placebo as the denominator, with two-sided 95% confidence interval

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence associated with the use of a drug in participants, whether or not considered drug related. An AE or suspected adverse reaction is considered serious (an SAE) if it is fatal, life-threatening, causes in-patient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect in a neonate/infant born to a mother or father exposed to study treatment or is an important medical event. Treatment-emergent adverse events are reported.
Time Frame: From first dose of study drug up to 28 days after last dose for each intervention (Up to approximately 4 Years)
Population: Safety Analysis Set (SAS) included all participants who received at least one dose of study drug (AG-120 or Placebo).
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo | After Crossover to AG-120
Number analyzed (Participants) | 123 | 59 | 43
percentage of participants
  AEs | 97.6 | 96.6 | 95.3
  SAEs | 35.0 | 23.7 | 27.9

3. Secondary Outcome: Percentage of Participants Who Experienced Laboratory Abnormalities Reported as Grade 3 or Higher Adverse Events
Description: The laboratory parameters evaluated by the investigator included hematology and chemistry. Laboratory abnormalities reported in this endpoint are Grade 3 or higher adverse events. Grading categories were determined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03.
Time Frame: From first dose of the study drug up to end of treatment visit for each intervention (Up to approximately 4 Years)
Population: SAS included all participants who received at least one dose of study drug (AG-120 or Placebo).
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo | After Crossover to AG-120
Number analyzed (Participants) | 123 | 59 | 43
percentage of participants
  Anaemia | 7.3 | 0.0 | 9.3
  Platelet Count Decreased | 2.4 | 0.0 | 2.3
  Neutrophil Count Decreased | 1.6 | 0.0 | 0.0
  White Blood Cell Count Decreased | 1.6 | 0.0 | 0.0
  Lymphocyte Count Decreased | 0.8 | 3.4 | 0.0
  Thrombocytopenia | 0.8 | 0.0 | 0.0
  Blood Loss Anaemia | 0.8 | 0.0 | 0.0
  Blood Bilirubin Increased | 5.7 | 1.7 | 7.0
  Hyponatraemia | 5.7 | 10.2 | 2.3
  Aspartate Aminotransferase Increased | 4.9 | 1.7 | 4.7
  Hypophosphataemia | 3.3 | 5.1 | 4.7
  Hyperbilirubinaemia | 3.3 | 0.0 | 0.0
  Hyperkalaemia | 2.4 | 3.4 | 2.3
  Blood Alkaline Phosphatase Increased | 2.4 | 5.1 | 0.0
  Alanine Aminotransferase Increased | 1.6 | 0.0 | 2.3
  Hypoalbuminaemia | 1.6 | 1.7 | 0.0
  Gamma-glutamyltransferase Increased | 0.8 | 1.7 | 0.0
  Hypercalcaemia | 0.8 | 1.7 | 0.0
  Hyperuricaemia | 0.8 | 0.0 | 0.0
  Hypokalaemia | 0.8 | 1.7 | 2.3
  Transaminases Increased | 0.8 | 0.0 | 0.0
  Blood Uric Acid Increased | 0.0 | 1.7 | 0.0

4. Secondary Outcome: Percentage of Participants With Clinically Significant Grade 3 or Higher Vital Signs AEs
Description: Clinically significant vital signs were recorded as adverse events; there were some vital signs reported as Grade 3 or higher adverse events. Grading categories were determined by NCI CTCAE, version 4.03.
Time Frame: From first dose of the study drug up to end of treatment visit for each intervention (Up to approximately 4 Years)
Population: SAS included all participants who received at least one dose of study drug (AG-120 or Placebo).
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo | After Crossover to AG-120
Number analyzed (Participants) | 123 | 59 | 43
percentage of participants
  Pyrexia | 0.8 | 0.0 | 2.3
  Weight Decreased | 0.8 | 1.7 | 0.0
  Hypertension | 1.6 | 1.7 | 7.0
  Hypotension | 1.6 | 1.7 | 2.3

5. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score classified participants according to their functional impairment, with scores ranging from 0 to 4. ECOG PS: 0 = fully active, able to carry on all pre-disease performance without restriction; 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work; 2 = ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3 = capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = completely disabled, cannot carry on any self-care, totally confined to bed or chair. A higher score means a worse functional status.
Time Frame: Baseline
Population: ITT population included all participants who were randomized, with the treatment group designated according to the randomization.
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 126 | 61
percentage of participants
  0 | 39.7 | 31.1
  1 | 59.5 | 67.2
  2 | 0.0 | 1.6
  3 | 0.8 | 0.0
  4 | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants Who Required At Least One Concomitant Medications During the Treatment
Description: Concomitant medications were medications that were ongoing or initiated after the first dose of the study drug but before the last dose plus 28 days. Percentage of participants who required at least one concomitant medications during the study along with their prescribed study drug (AG-120 or placebo) were reported.
Time Frame: From first dose of study drug up to 28 days after last dose (Up to approximately 4 Years)
Population: SAS included all participants who received at least one dose of study drug (AG-120 or Placebo).
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo | After Crossover to AG-120
Number analyzed (Participants) | 123 | 59 | 43
percentage of participants | 99.2 | 98.3 | 95.3

7. Secondary Outcome: Percentage of Participants With Abnormal Electrocardiogram (ECG) Changes Reported as Adverse Events
Time Frame: Pre-dose C1D1, C2D1; Post-dose C1D1, C1D15, C2D1 and Day 1 of C3D1 and all cycles thereafter up to last dose plus 28 days (Up to approximately 4 years)
Population: SAS included all participants who received at least one dose of study drug (AG-120 or Placebo).
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo | After Crossover to AG-120
Number analyzed (Participants) | 123 | 59 | 43
percentage of participants
  Electrocardiogram QT Prolonged | 9.8 | 3.4 | 2.3
  Electrocardiogram Abnormal | 0.8 | 0.0 | 0.0

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time in months from date of randomization to the date of death due to any cause. Participants without documentation of death at the time of the final collection were censored at the date the participant was last known to be alive, or the final collection date, whichever is earlier.
Time Frame: From date of randomization until the date of death due to any cause (Up to approximately 2 years)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 126 | 61
months | 10.3 [7.8 to 12.4] | 7.5 [4.8 to 11.1]
Statistical Analysis 1: Comparison: AG-120 vs Placebo; Test type: Superiority; p = 0.093, Log Rank — P-value was calculated from the one-sided stratified log-rank test. Stratification factor was the number of prior line of therapies at randomization; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.56 to 1.12] — Hazard ratio was calculated from the stratified Cox regression model with placebo as the comparator, with two-sided 95% CI. Stratification factor was the number of prior line of therapies at randomization

9. Secondary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator RECIST Version 1.1
Description: ORR as assessed by the investigator was defined as the percentage of participants with a best overall response (BOR) defined as complete response (CR) or partial response (PR) per RECIST v1.1. CR: disappearance of all target and non-target lesions (TLs) and all pathological lymph nodes (LNs) (target and non target), with short axis <10mm. PR: ≥30% decrease in sum of diameters (SOD) from Baseline.
Time Frame: From the date of randomization up to confirmed CR or PR (Up to approximately 2 years)
Population: ITT population included all participants who were randomized, with the treatment group designated according to the randomization. Number analyzed is the number of participants with data available for analyses at the specified time point. Two participants were excluded from the analysis as they were randomized in the study after the data cutoff date (31 January 2019) for the analysis of tumor response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 124 | 61
percentage of participants | 3.2 [0.9 to 8.1] | 1.6 [0.0 to 8.8]
Statistical Analysis 1: Comparison: AG-120 vs Placebo; Test type: Superiority; p = 0.466, Fisher Exact — P-value was calculated from 1-sided Fisher exact test

10. Secondary Outcome: ORR as Assessed by the IRC Per RECIST v1.1
Description: ORR as assessed by the IRC was defined as the percentage of participants with a best overall response (BOR) defined as complete response (CR) or partial response (PR) per RECIST v1.1. CR: disappearance of all target and non-target lesions (TLs) and all pathological lymph nodes (LNs) (target and non target), with short axis <10mm. PR: ≥30% decrease in sum of diameters (SOD) from Baseline.
Time Frame: From the date of randomization up to confirmed CR or PR (Up to approximately 2 years)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 124 | 61
percentage of participants | 2.4 [0.5 to 6.9] | 0 [0.0 to 5.9]
Statistical Analysis 1: Comparison: AG-120 vs Placebo; Test type: Superiority; p = 0.299, Fisher Exact — P-value was calculated from 1-sided Fisher exact test

11. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator
Description: DOR was defined as the time in months from date of first documented CR or PR to date of first documented disease progression or death due to any cause, whichever is earlier, as assessed by the Investigator per RECIST v1.1. CR: disappearance of all target and non-target lesions (TLs) and all pathological lymph nodes (LNs) (target and non target), with short axis <10mm. PR: ≥30% decrease in sum of diameters (SOD) from Baseline. Participants with response and without progression were censored at the last observation.
Time Frame: From the date of first confirmed CR or PR to disease progression or death regardless of cause (Up to approximately 2 years)
Population: Participants with CR or PR per investigator assessment by the data cutoff date (31 January 2019) for the analysis of tumor response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 4 | 1
months | NA [NA to NA] — Median, lower limit and upper limit were not available due to the insufficient number of participants with events. | NA [NA to NA] — Median, lower limit and upper limit were not available due to the insufficient number of participants with events.

12. Secondary Outcome: DOR as Assessed by the IRC Per RECIST v1.1
Description: DOR was defined as the time in months from date of first documented CR or PR to date of first documented disease progression or death due to any cause, whichever is earlier, as assessed by the IRC per RECIST v1.1. CR: disappearance of all target and non-target lesions (TLs) and all pathological lymph nodes (LNs) (target and non target), with short axis <10mm. PR: ≥30% decrease in sum of diameters (SOD) from Baseline. Participants with response and without progression were censored at the last observation.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 3 | 0
months | NA [NA to NA] — Median, lower limit and upper limit were not available due to the insufficient number of participants with events. |

13. Secondary Outcome: Time to Response (TTR) as Assessed by the Investigator
Description: TTR was defined as the time from date of randomization to date of first documented CR or PR for responders, as assessed by the Investigator per RECIST v1.1. CR: disappearance of all target and non-target lesions (TLs) and all pathological lymph nodes (LNs) (target and non target), with short axis <10mm. PR: ≥30% decrease in sum of diameters (SOD) from Baseline. Only responders were analyzed for this outcome measure.
Time Frame: From the date of randomization up to the date of first documented CR or PR (Up to approximately 2 years)
Population: Participants with CR or PR per investigator assessment by the data cutoff date (31 January 2019) were analyzed for tumor response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 4 | 1
months | NA [NA to NA] — Median, upper and lower limit were not available due to the insufficient number of participants with events. | NA [NA to NA] — Median, upper and lower limit were not available due to the insufficient number of participants with events.

14. Secondary Outcome: TTR as Assessed by the IRC Per RECIST v1.1
Description: TTR was defined as the time from date of randomization to date of first documented CR or PR for responders, as assessed by the IRC per RECIST v1.1. CR: disappearance of all target and non-target lesions (TLs) and all pathological lymph nodes (LNs) (target and non target), with short axis <10mm. PR: ≥30% decrease in sum of diameters (SOD) from Baseline. Only responders were analyzed for this outcome measure.
Time Frame: From the date of randomization up to the date of first documented CR or PR (Up to approximately 2 years)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 3 | 0
months | NA [NA to NA] — Median, upper and lower limit were not available due to the insufficient number of participants with events. |

15. Secondary Outcome: PFS as Determined by Investigator
Description: PFS was defined as the time from date of randomization to the date of first documented disease progression as assessed by the investigator using RECIST v1.1, or date of death due to any cause, whichever occurred first. Disease progression was defined as ≥20% increase in sum of the diameter of target lesions, taking as reference the smallest sum diameter recorded since the treatment started. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm or the appearance of 1 or more new lesions. No progression or death by data cutoff date was censored at the last adequate assessment date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 124 | 61
months | 2.7 [1.6 to 3.6] | 1.4 [1.4 to 2.5]
Statistical Analysis 1: Comparison: AG-120 vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — P-value was calculated from one-sided stratified log-rank test. Stratification factor was the number of prior line of therapies at randomization; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.33 to 0.68] — Hazard ratio was calculated from the stratified Cox regression model with placebo as the denominator, with two-sided 95% CI. Stratification factor was the number of prior line of therapies at randomization

16. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQOL) Based on European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire- Core 30 Subscales Scores
Description: EORTC-QLQ-C30 is the European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire - Core Questionnaire. For EORTC QLQ-C30, subscales of physical functioning, pain, and appetite loss were assessed. These had 4 response levels (not at all, a little, quite a bit, and very much). For functional scales, higher scores=better QOL (positive change from Baseline=improvement). For symptom scales, lower scores=better QOL (negative change from Baseline=improvement). Using linear transformation, raw scores were standardized, so that scores ranged from 0 to 100.
Time Frame: Cycle 2 Day 1 and Cycle 3 Day 1
Population: ITT population included all randomized participants, with treatment group designated according to the randomization. Overall Number of Participants Analyzed is the number of participants with data available for analyses at baseline and the given post-baseline timepoints. Number Analyzed at a particular timepoint is the number of participants with data available for analyses at baseline and given timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 73 | 23
score on a scale
  Cycle 2 Day 1: Physical Functioning: number analyzed (Participants) | 67 | 21
  Cycle 2 Day 1: Physical Functioning | -2.4 (1.75) | -13.3 (2.95)
  Cycle 2 Day 1: Pain: number analyzed (Participants) | 67 | 21
  Cycle 2 Day 1: Pain | 2.2 (2.48) | 12.5 (4.35)
  Cycle 2 Day 1: Appetite Loss: number analyzed (Participants) | 67 | 21
  Cycle 2 Day 1: Appetite Loss | 7.9 (2.60) | 4.3 (4.55)
  Cycle 3 Day 1: Physical Functioning: number analyzed (Participants) | 50 | 9
  Cycle 3 Day 1: Physical Functioning | -0.2 (1.89) | -12.6 (3.88)
  Cycle 3 Day 1: Pain: number analyzed (Participants) | 50 | 9
  Cycle 3 Day 1: Pain | -1.2 (2.73) | -5.3 (5.96)
  Cycle 3 Day 1: Appetite Loss: number analyzed (Participants) | 50 | 9
  Cycle 3 Day 1: Appetite Loss | -0.5 (2.89) | 3.2 (6.40)
Statistical Analysis 1: Comparison: AG-120 vs Placebo; Cycle 2 Day 1: Physical Functioning; Test type: Other; Least-squares mean difference = 11.0, 95% CI 2-sided [4.23 to 17.73]
Statistical Analysis 2: Comparison: AG-120 vs Placebo; Cycle 2 Day 1: Pain; Test type: Other; Least-squares mean difference = -10.4, 95% CI 2-sided [-20.18 to -0.52]
Statistical Analysis 3: Comparison: AG-120 vs Placebo; Cycle 2 Day 1: Appetite Loss; Test type: Other; Least-squares mean difference = 3.6, 95% CI 2-sided [-6.65 to 13.91]
Statistical Analysis 4: Comparison: AG-120 vs Placebo; Cycle 3 Day 1: Physical Functioning; Test type: Other; Least-squares mean difference = 12.3, 95% CI 2-sided [3.85 to 20.78]
Statistical Analysis 5: Comparison: AG-120 vs Placebo; Cycle 3 Day 1: Pain; Test type: Other; Least-squares mean difference = 4.1, 95% CI 2-sided [-8.74 to 17.04]
Statistical Analysis 6: Comparison: AG-120 vs Placebo; Cycle 3 Day 1: Appetite Loss; Test type: Other; Least-squares mean difference = -3.7, 95% CI 2-sided [-17.46 to 10.11]

17. Secondary Outcome: Change From Baseline in HRQOL Based on: Quality of Life Questionnaire - Cholangiocarcinoma and Gallbladder Cancer Module (QLQ-BIL21)
Description: For HRQOL based on QLQ-BIL21, subscales of eating symptoms and pain symptoms were assessed. Each item is a 4-point Likert scale. There are 4 response levels (not at all, a little, quite a bit, and very much). Raw scores are converted into scale scores ranging from 0 to 100. For symptom scales, lower scores=better QOL (negative change from Baseline=improvement).
Time Frame: Cycle 2 Day 1 and Cycle 3 Day 1
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 70 | 22
score on a scale
  Cycle 2 Day 1: Pain: number analyzed (Participants) | 65 | 20
  Cycle 2 Day 1: Pain | 5.1 (1.94) | 10.1 (3.49)
  Cycle 2 Day 1: Appetite Loss: number analyzed (Participants) | 65 | 20
  Cycle 2 Day 1: Appetite Loss | 4.3 (1.84) | 3.6 (3.19)
  Cycle 3 Day 1: Pain: number analyzed (Participants) | 48 | 9
  Cycle 3 Day 1: Pain | 2.3 (2.16) | -2.1 (4.70)
  Cycle 3 Day 1: Appetite Loss: number analyzed (Participants) | 48 | 9
  Cycle 3 Day 1: Appetite Loss | -2.0 (2.02) | 4.1 (4.24)
Statistical Analysis 1: Comparison: AG-120 vs Placebo; Cycle 2 Day 1: Pain; Test type: Other; Least-squares mean difference = -5.1, 95% CI 2-sided [-12.93 to 2.80]
Statistical Analysis 2: Comparison: AG-120 vs Placebo; Cycle 2 Day 1: Appetite Loss; Test type: Other; Least-squares mean difference = 0.7, 95% CI 2-sided [-6.56 to 7.88]
Statistical Analysis 3: Comparison: AG-120 vs Placebo; Cycle 3 Day 1: Pain; Test type: Other; Least-squares mean difference = 4.4, 95% CI 2-sided [-5.82 to 14.55]
Statistical Analysis 4: Comparison: AG-120 vs Placebo; Cycle 3 Day 1: Appetite Loss; Test type: Other; Least-squares mean difference = -6.1, 95% CI 2-sided [-15.34 to 3.12]

18. Secondary Outcome: Percentage of Participants With Change Based on HRQOL: Patient Global Impression of Change (PGI-C)
Description: The PGI-C is a self-rated evaluative instrument for assessment across 3 domains (physical function, appetite loss, and pain). The PGI-C is measured using a 7-point Likert scale, with 6= very much better, 5= moderately better, 4= a little better, 3= no change, 2= a little worse, 1= moderately worse, and 0= very much worse. A lower score indicates a worse outcome. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Cycle 2 Day 1 and Cycle 3 Day 1
Population: ITT population included all participants who were randomized, with the treatment group designated according to the randomization. Overall number analyzed is the number of participants available for analysis. Number analyzed is the number of participants available for analysis at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 67 | 22
percentage of participants
  Physical Change: Cycle 2 Day 1: Very Much Worse | 1.5 | 0.0
  Physical Change: Cycle 2 Day 1: Moderately Worse | 4.5 | 13.6
  Physical Change: Cycle 2 Day 1: A Little Worse | 22.4 | 9.1
  Physical Change: Cycle 2 Day 1: No Change | 38.8 | 27.3
  Physical Change: Cycle 2 Day 1: A Little Better | 22.4 | 36.4
  Physical Change: Cycle 2 Day 1: Moderately Better | 9.0 | 9.1
  Physical Change: Cycle 2 Day 1: Very Much Better | 1.5 | 4.5
  Physical Change: Cycle 3 Day 1: Very Much Worse: number analyzed (Participants) | 51 | 12
  Physical Change: Cycle 3 Day 1: Very Much Worse | 2.0 | 0.0
  Physical Change: Cycle 3 Day 1: Moderately Worse: number analyzed (Participants) | 51 | 12
  Physical Change: Cycle 3 Day 1: Moderately Worse | 5.9 | 0.0
  Physical Change: Cycle 3 Day 1: A Little Worse: number analyzed (Participants) | 51 | 12
  Physical Change: Cycle 3 Day 1: A Little Worse | 3.9 | 8.3
  Physical Change: Cycle 3 Day 1: No Change: number analyzed (Participants) | 51 | 12
  Physical Change: Cycle 3 Day 1: No Change | 41.2 | 58.3
  Physical Change: Cycle 3 Day 1: A Little Better: number analyzed (Participants) | 51 | 12
  Physical Change: Cycle 3 Day 1: A Little Better | 29.4 | 16.7
  Physical Change: Cycle 3 Day 1: Moderately Better: number analyzed (Participants) | 51 | 12
  Physical Change: Cycle 3 Day 1: Moderately Better | 15.7 | 16.7
  Physical Change: Cycle 3 Day 1: Very Much Better: number analyzed (Participants) | 51 | 12
  Physical Change: Cycle 3 Day 1: Very Much Better | 2.0 | 0.0
  Appetite Change: Cycle 2 Day 1: Very Much Worse | 1.5 | 0.0
  Appetite Change: Cycle 2 Day 1: Moderately Worse | 4.5 | 4.5
  Appetite Change: Cycle 2 Day 1: A Little Worse | 20.9 | 18.2
  Appetite Change: Cycle 2 Day 1: No Change | 50.7 | 45.5
  Appetite Change: Cycle 2 Day 1: A Little Better | 13.4 | 13.6
  Appetite Change: Cycle 2 Day 1: Moderately Better | 7.5 | 9.1
  Appetite Change: Cycle 2 Day 1: Very Much Better | 1.5 | 9.1
  Appetite Change: Cycle 3 Day 1: Very Much Worse: number analyzed (Participants) | 51 | 12
  Appetite Change: Cycle 3 Day 1: Very Much Worse | 0.0 | 0.0
  Appetite Change: Cycle 3 Day 1: Moderately Worse: number analyzed (Participants) | 51 | 12
  Appetite Change: Cycle 3 Day 1: Moderately Worse | 5.9 | 8.3
  Appetite Change: Cycle 3 Day 1: A Little Worse: number analyzed (Participants) | 51 | 12
  Appetite Change: Cycle 3 Day 1: A Little Worse | 5.9 | 0.0
  Appetite Change: Cycle 3 Day 1: No Change: number analyzed (Participants) | 51 | 12
  Appetite Change: Cycle 3 Day 1: No Change | 64.7 | 50.0
  Appetite Change: Cycle 3 Day 1: A Little Better: number analyzed (Participants) | 51 | 12
  Appetite Change: Cycle 3 Day 1: A Little Better | 11.8 | 25.0
  Appetite Change: Cycle 3 Day 1: Moderately Better: number analyzed (Participants) | 51 | 12
  Appetite Change: Cycle 3 Day 1: Moderately Better | 7.8 | 0.0
  Appetite Change: Cycle 3 Day 1: Very Much Better: number analyzed (Participants) | 51 | 12
  Appetite Change: Cycle 3 Day 1: Very Much Better | 3.9 | 16.7
  Pain Change: Cycle 2 Day 1: Very Much Worse | 0.0 | 0.0
  Pain Change: Cycle 2 Day 1: Moderately Worse | 9.0 | 13.6
  Pain Change: Cycle 2 Day 1: A Little Worse | 9.0 | 9.1
  Pain Change: Cycle 2 Day 1: No Change | 64.2 | 54.5
  Pain Change: Cycle 2 Day 1: A Little Better | 7.5 | 18.2
  Pain Change: Cycle 2 Day 1: Moderately Better | 10.4 | 4.5
  Pain Change: Cycle 2 Day 1: Very Much Better | 0.0 | 0.0
  Pain Change: Cycle 3 Day 1: Very Much Worse: number analyzed (Participants) | 51 | 12
  Pain Change: Cycle 3 Day 1: Very Much Worse | 0.0 | 0.0
  Pain Change: Cycle 3 Day 1: Moderately Worse: number analyzed (Participants) | 51 | 12
  Pain Change: Cycle 3 Day 1: Moderately Worse | 3.9 | 0.0
  Pain Change: Cycle 3 Day 1: A Little Worse: number analyzed (Participants) | 51 | 12
  Pain Change: Cycle 3 Day 1: A Little Worse | 11.8 | 8.3
  Pain Change: Cycle 3 Day 1: No Change: number analyzed (Participants) | 51 | 12
  Pain Change: Cycle 3 Day 1: No Change | 60.8 | 66.7
  Pain Change: Cycle 3 Day 1: A Little Better: number analyzed (Participants) | 51 | 12
  Pain Change: Cycle 3 Day 1: A Little Better | 7.8 | 8.3
  Pain Change: Cycle 3 Day 1: Moderately Better: number analyzed (Participants) | 51 | 12
  Pain Change: Cycle 3 Day 1: Moderately Better | 11.8 | 8.3
  Pain Change: Cycle 3 Day 1: Very Much Better: number analyzed (Participants) | 51 | 12
  Pain Change: Cycle 3 Day 1: Very Much Better | 3.9 | 8.3

19. Secondary Outcome: Percentage of Participants With Severity Based on HRQOL: Patient Global Impression of Severity (PGI-S)
Description: The anchor-based questionnaire PGI-S contains the following 3 items (the severity of the physical functioning decline over the past week, the severity of the appetite decrease over the past week, and the severity of the pain over the past week). The PGI-S was measured using the possible outcomes none, mild, moderate, severe, and very severe. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Cycle 2 Day 1 and Cycle 3 Day 1
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 67 | 22
percentage of participants
  Physical Decline: Cycle 2 Day 1: None | 55.2 | 31.8
  Physical Decline: Cycle 2 Day 1: Mild | 23.9 | 27.3
  Physical Decline: Cycle 2 Day 1: Moderate | 16.4 | 31.8
  Physical Decline: Cycle 2 Day 1: Severe | 3.0 | 9.1
  Physical Decline: Cycle 2 Day 1: Very Severe | 1.5 | 0.0
  Physical Decline: Cycle 3 Day 1: None: number analyzed (Participants) | 51 | 12
  Physical Decline: Cycle 3 Day 1: None | 70.6 | 75.0
  Physical Decline: Cycle 3 Day 1: Mild: number analyzed (Participants) | 51 | 12
  Physical Decline: Cycle 3 Day 1: Mild | 11.8 | 16.7
  Physical Decline: Cycle 3 Day 1: Moderate: number analyzed (Participants) | 51 | 12
  Physical Decline: Cycle 3 Day 1: Moderate | 15.7 | 8.3
  Physical Decline: Cycle 3 Day 1: Severe: number analyzed (Participants) | 51 | 12
  Physical Decline: Cycle 3 Day 1: Severe | 2.0 | 0.0
  Physical Decline: Cycle 3 Day 1: very Severe: number analyzed (Participants) | 51 | 12
  Physical Decline: Cycle 3 Day 1: very Severe | 0.0 | 0.0
  Appetite Decrease: Cycle 2 Day 1: None | 53.7 | 45.5
  Appetite Decrease: Cycle 2 Day 1: Mild | 32.8 | 13.6
  Appetite Decrease: Cycle 2 Day 1: Moderate | 10.4 | 36.4
  Appetite Decrease: Cycle 2 Day 1: Severe | 1.5 | 4.5
  Appetite Decrease: Cycle 2 Day 1: Very Severe | 1.5 | 0.0
  Appetite Decrease: Cycle 3 Day 1: None: number analyzed (Participants) | 51 | 12
  Appetite Decrease: Cycle 3 Day 1: None | 70.6 | 58.3
  Appetite Decrease: Cycle 3 Day 1: Mild: number analyzed (Participants) | 51 | 12
  Appetite Decrease: Cycle 3 Day 1: Mild | 15.7 | 25.0
  Appetite Decrease: Cycle 3 Day 1: Moderate: number analyzed (Participants) | 51 | 12
  Appetite Decrease: Cycle 3 Day 1: Moderate | 7.8 | 16.7
  Appetite Decrease: Cycle 3 Day 1: Severe: number analyzed (Participants) | 51 | 12
  Appetite Decrease: Cycle 3 Day 1: Severe | 5.9 | 0.0
  Appetite Decrease: Cycle 3 Day 1: Very Severe: number analyzed (Participants) | 51 | 12
  Appetite Decrease: Cycle 3 Day 1: Very Severe | 0.0 | 0.0
  Pain Severity: Cycle 2 Day 1: None | 32.8 | 31.8
  Pain Severity: Cycle 2 Day 1: Mild | 38.8 | 13.6
  Pain Severity: Cycle 2 Day 1: Moderate | 23.9 | 40.9
  Pain Severity: Cycle 2 Day 1: Severe | 4.5 | 9.1
  Pain Severity: Cycle 2 Day 1: Very Severe | 0.0 | 4.5
  Pain Severity: Cycle 3 Day 1: None: number analyzed (Participants) | 51 | 12
  Pain Severity: Cycle 3 Day 1: None | 39.2 | 33.3
  Pain Severity: Cycle 3 Day 1: Mild: number analyzed (Participants) | 51 | 12
  Pain Severity: Cycle 3 Day 1: Mild | 35.3 | 25.0
  Pain Severity: Cycle 3 Day 1: Moderate: number analyzed (Participants) | 51 | 12
  Pain Severity: Cycle 3 Day 1: Moderate | 17.6 | 41.7
  Pain Severity: Cycle 3 Day 1: Severe: number analyzed (Participants) | 51 | 12
  Pain Severity: Cycle 3 Day 1: Severe | 7.8 | 0.0
  Pain Severity: Cycle 3 Day 1: Very Severe: number analyzed (Participants) | 51 | 12
  Pain Severity: Cycle 3 Day 1: Very Severe | 0.0 | 0.0

20. Secondary Outcome: Percentage of Participants With Each EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) Dimension Response
Description: The EQ-5D-5L assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Cycle 3 Day 1
Population: ITT population included all participants who were randomized, with the treatment group designated according to the randomization. Overall number analyzed is the number of participants available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 50 | 12
percentage of participants
  Mobility: No Problems Walking | 52.0 | 41.7
  Mobility: Slight Problems Walking | 28.0 | 25.0
  Mobility: Moderate Problems Walking | 16.0 | 33.3
  Mobility: Severe Problems Walking | 4.0 | 0.0
  Mobility: Unable to Walk | 0.0 | 0.0
  Self-Care: No Problems Washing or Dressing | 88.0 | 83.3
  Self-Care: Slight Problems Washing or Dressing | 8.0 | 16.7
  Self-Care: Moderate Problems Washing or Dressing | 2.0 | 0.0
  Self-Care: Severe Problems Washing or Dressing | 2.0 | 0.0
  Usual Activities: No Problems Doing Usual Activities | 42.0 | 33.3
  Usual Activities: Slight Problems Doing Usual Activities | 34.0 | 41.7
  Usual Activities: Moderate Problems Doing Usual Activities | 16.0 | 25.0
  Usual Activities: Severe Problems Doing Usual Activities | 8.0 | 0.0
  Usual Activities: Unable to do Usual Activities | 0.0 | 0.0
  Pain/Discomfort: No Pain or Discomfort | 40.0 | 41.7
  Pain/Discomfort: Slight Pain or Discomfort | 42.0 | 33.3
  Pain/Discomfort: Moderate Pain or Discomfort | 10.0 | 25.0
  Pain/Discomfort: Severe Pain or Discomfort | 6.0 | 0.0
  Pain/Discomfort: Extreme Pain or Discomfort | 2.0 | 0.0
  Anxiety/Depression: Not Anxious or Depressed | 50.0 | 33.3
  Anxiety/Depression: Slightly Anxious or Depressed | 44.0 | 33.3
  Anxiety/Depression: Moderately Anxious or Depressed | 6.0 | 25.0
  Anxiety/Depression: Severely Anxious or Depressed | 0.0 | 8.3

21. Secondary Outcome: Change From Baseline in EQ-5D-5L Visual Analogue Scale (EQ-5D-5L VAS) Score
Description: The EQ visual analogue scale records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine." Responses are marked on a 0-100 scale with higher scores indicating higher health-related quality of life (i.e., better outcome).
Time Frame: Cycle 3 Day 1
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AG-120 | Placebo
Number analyzed (Participants) | 46 | 9
score on a scale | 4.6 (13.48) | -2.8 (7.76)

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of AG-120
Description: Crossover C1D1 and crossover C2D1 visits were combined with C1D1 and C2D1 visits, respectively for the analysis of this endpoint.
Time Frame: Post-dose Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle = 28 days)
Population: Pharmacokinetic (PK) Analysis Population consisted of all participants who were enrolled and received at least one dose of study medication (AG-120) with sufficient plasma sample data to assess PK parameters. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Randomization Phase AG-120 Plus Cross Over Phase AG-120: Participants received AG-120 500 mg, tablet, orally, QD in each 28-day treatment cycle, until occurrence of disease progression, unacceptable toxicity, confirmed pregnancy, death, subject withdrawal, lost to follow-up, or the sponsor ended the study. Participants who experienced disease progression and received placebo were allowed to cross over to receive AG-120 500 mg, tablet, orally, QD in each 28-day treatment cycle.
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 142
ng/mL
  Cycle 1 Day 1 | 4424.0 (1808.07)
  Cycle 2 Day 1: number analyzed (Participants) | 107
  Cycle 2 Day 1 | 5050.5 (1666.07)

23. Secondary Outcome: Time to Reach Maximal Plasma Concentration (Tmax) of AG-120
Description: as for outcome 22
Time Frame: Post-dose Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle = 28 days)
Population: PK Analysis Population consisted of all participants who were enrolled and received at least one dose of study medication (AG-120) with sufficient plasma sample data to assess PK parameters. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 142
hours (h)
  Cycle 1 Day 1 | 2.63 [0.50 to 4.87]
  Cycle 2 Day 1: number analyzed (Participants) | 107
  Cycle 2 Day 1 | 2.07 [0.50 to 4.08]

24. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC0-24)
Description: Crossover C2D1 visit was combined with C2D1 visit for the analysis of this endpoint.
Time Frame: Post-dose of Cycle 2 Day 1 (each cycle = 28 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 107
h*ng/mL | 91219.4 (31574.57)

25. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 4 Hours (AUC0-4)
Description: as for outcome 22
Time Frame: Post-dose of Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle = 28 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 141
h*ng/mL
  Cycle 1 Day 1 | 10972.2 (5044.1)
  Cycle 2 Day 1: number analyzed (Participants) | 106
  Cycle 2 Day 1 | 16651.7 (5269.9)

26. Secondary Outcome: Accumulation Ratio Based on AUC0-4 (Racc AUC0-4)
Description: Crossover C2D1 visit was combined with C2D1 visit for the analysis of this endpoint.
Time Frame: Post-dose Cycle 2 Day 1 (each cycle = 28 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 98
ratio | 1.6881 (0.83303)

27. Secondary Outcome: Accumulation Ratio Based on Cmax (Racc Cmax)
Description: Crossover C2D1 visit was combined with C2D1 visit for the analysis of this endpoint.
Time Frame: Post-dose Cycle 2 Day 1 (each cycle = 28 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 100
ratio | 1.2369 (0.50798)

28. Secondary Outcome: Plasma 2-hydroxyglutarate (2-HG) Levels of AG-120: B (Baseline Effect Value)
Description: B is the Baseline Effect Value. Crossover C1D1 and crossover C2D1 visits were combined with C1D1 and C2D1 visits, respectively for the analysis of this endpoint.
Time Frame: Post-dose Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle = 28 days)
Population: Pharmacodynamic (PD) Analysis Population consisted of all participants who were enrolled and received any dose of study medication (AG-120) with sufficient plasma sample data to assess pharmacodynamic parameters. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 142
ng/mL
  Cycle 1 Day 1 | 1107.70 (1709.919)
  Cycle 2 Day 1: number analyzed (Participants) | 108
  Cycle 2 Day 1 | 795.09 (938.677)

29. Secondary Outcome: Plasma 2-hydroxyglutarate (2-HG) Levels of AG-120: AUEC0-4
Description: AUEC0-4 is the area of the response curve from time point zero (predose) up to 4 hr postdose. Crossover C1D1 and crossover C2D1 visits were combined with C1D1 and C2D1 visits, respectively for the analysis of this endpoint.
Time Frame: Post-dose Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle = 28 days)
Population: PD Analysis Population consisted of all participants who were enrolled and received any dose of study medication (AG-120) with sufficient plasma sample data to assess pharmacodynamic parameters. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 141
h*ng/mL
  Cycle 1 Day 1 | 3334.3 (4785.48)
  Cycle 2 Day 1: number analyzed (Participants) | 107
  Cycle 2 Day 1 | 368.4 (278.78)

30. Secondary Outcome: Plasma 2-hydroxyglutarate (2-HG) Levels of AG-120: %BAUEC0-4
Description: %BAUEC0-4 is the percent inhibition for AUEC0-4. Crossover C1D1 and crossover C2D1 visits were combined with C1D1 and C2D1 visits, respectively for the analysis of this endpoint.
Time Frame: Post-dose Cycle 1 Day 1 and Cycle 2 Day 1 (each cycle = 28 days)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 141
percent
  Cycle 1 Day 1 | 20.22090 (10.13659)
  Cycle 2 Day 1: number analyzed (Participants) | 107
  Cycle 2 Day 1 | 74.9750 (22.53852)

31. Secondary Outcome: Plasma 2-hydroxyglutarate (2-HG) Levels of AG-120: Rtrough
Description: Rtrough is the observed response value at the end of a dosing interval. Crossover C2D1 visit was combined with C2D1 visit for the analysis of this endpoint.
Time Frame: Post-dose Cycle 2 Day 1 (each cycle = 28 days)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 108
ng/mL | 97.66 (72.838)

32. Secondary Outcome: Plasma 2-hydroxyglutarate (2-HG) Levels of AG-120: %BRtrough
Description: %BRtrough is the percent inhibition for Rtrough. Crossover C2D1 visit was combined with C2D1 visit for the analysis of this endpoint.
Time Frame: Post-dose Cycle 2 Day 1 (each cycle = 28 days)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Randomization Phase AG-120 Plus Cross Over Phase AG-120
Number analyzed (Participants) | 108
percent | 73.726 (23.3113)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after last dose for each intervention (Up to approximately 4 years)
Description: All-Cause Mortality was assessed as per ITT population. Adverse Events: Safety Analysis Set included all participants who received at least one dose of study treatment.
Arm/Group | AG-120 | Placebo | After Cross Over to AG-120
All-Cause Mortality (participants affected / at risk) | 99/126 | 14/61 | 34/43
Serious Adverse Events (participants affected / at risk) | 43/123 | 14/59 | 12/43
Other Adverse Events (participants affected / at risk) | 118/123 | 56/59 | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-120 (N=123) | Placebo (N=59) | After Cross Over to AG-120 (N=43)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 3 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 0
Sepsis (Infections and infestations) | 4 | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Thecal sac compression (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AG-120 (N=123) | Placebo (N=59) | After Cross Over to AG-120 (N=43)
Nausea (Gastrointestinal disorders) | 52 | 17 | 12
Diarrhoea (Gastrointestinal disorders) | 43 | 10 | 12
Fatigue (General disorders) | 38 | 10 | 10
Abdominal pain (Gastrointestinal disorders) | 30 | 9 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 5 | 5
Decreased appetite (Metabolism and nutrition disorders) | 30 | 11 | 6
Ascites (Gastrointestinal disorders) | 25 | 7 | 5
Vomiting (Gastrointestinal disorders) | 28 | 11 | 5
Anaemia (Blood and lymphatic system disorders) | 23 | 3 | 7
Oedema peripheral (General disorders) | 17 | 6 | 9
Constipation (Gastrointestinal disorders) | 20 | 11 | 5
Asthenia (General disorders) | 17 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 7 | 2
Pyrexia (General disorders) | 16 | 6 | 2
Headache (Nervous system disorders) | 16 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 13 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 10 | 4
Abdominal distension (Gastrointestinal disorders) | 13 | 5 | 2
Blood alkaline phosphatase increased (Investigations) | 11 | 6 | 4
Blood bilirubin increased (Investigations) | 12 | 4 | 2
Hypertension (Vascular disorders) | 11 | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 6 | 1
Weight decreased (Investigations) | 10 | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 10 | 2 | 4
Alanine aminotransferase increased (Investigations) | 11 | 1 | 3
Insomnia (Psychiatric disorders) | 12 | 3 | 3
Electrocardiogram QT prolonged (Investigations) | 11 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 6 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 10 | 0 | 2
Dizziness (Nervous system disorders) | 7 | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 4 | 3
White blood cell count decreased (Investigations) | 9 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3 | 3
Chills (General disorders) | 8 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 3 | 3
Blood creatinine increased (Investigations) | 7 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 8 | 0 | 0
Urinary tract infection (Infections and infestations) | 7 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0 | 3
Confusional state (Psychiatric disorders) | 4 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 7 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 1
Gait disturbance (General disorders) | 0 | 3 | 0
Platelet count decreased (Investigations) | 7 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained from the clinical study will be used towards the development of ivosidenib and may be disclosed to regulatory authority(ies), other Investigators, corporate partners, or consultants as required.

DOCUMENTS (3):
  • Study Protocol: Protocol v6 (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT02989857/Prot_000.pdf
  • Study Protocol: Protocol v7 (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT02989857/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT02989857/SAP_001.pdf